CLINICAL TRIAL: NCT06962397
Title: Research on the Effectiveness of the Method of Active Examination of Artificially Simulated Textures Generated by Programmable Transcutaneous Electrical Stimulation as a Method of Restoring Sensorimotor Function of the Upper Limbs
Brief Title: Effectiveness of Active Exploration of Simulated Textures for Sensorimotor Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Center of Cerebrovascular Pathology and Stroke, Russian Federation Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ActiveTouch01
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Sensorimotor Impairment Affecting the Upper Limb; Sensory Deficit; Rehabilitation; Tactile Disorders
Keywords: Stroke; Sensorimotor rehabilitation; Tactile stimulation; Upper limb recovery; Electrical stimulation; Virtual textures; Sensory training; Neurorehabilitation; Post-stroke therapy; Active touch paradigm; Functional electrical stimulation; Proprioception; Touch sensitivity; Stroke rehabilitation technology
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: This is a parallel-group, controlled trial. Participants are randomized into two groups. The experimental group receives 10 sessions of active sensory training using programmable electrical stimulation during virtual texture exploration, in addition to standard rehabilitation. The control group receives standard rehabilitation only. Both groups are evaluated pre- and post-intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Touch Sensory Training Intervention (Experimental): Participants in this arm undergo a novel sensory rehabilitation protocol based on the Active Touch Paradigm. This intervention integrates real-time functional electrical stimulation with voluntary finger movement across a touch-sensitive screen to explore virtual textures of varying densities. Each time a participant's finger crosses an invisible virtual grating line, a tactile sensation is delivered via electrical stimulation to the index finger. The system records finger trajectory, response time, and decision-making accuracy, offering real-time visual and tactile feedback to enhance sensory discrimination and neuroplasticity. The training consists of 180 trials divided into six blocks with breaks in between, and assessments are conducted before and after the intervention using tools such as the Touch-Test monofilament, Fugl-Meyer Assessment, and ARAT. This arm aims to evaluate the efficacy of active engagement and sensorimotor integration in promoting sensory recovery after stroke.
  Interventions: Device: Active Touch-Based Sensory Training
- Standard Rehabilitation Without Sensory Training (No Intervention): Participants in this arm receive standard post-stroke rehabilitation as prescribed by their physicians but do not undergo any form of targeted sensory training or participate in the Active Touch Paradigm. They complete the same pre- and post-intervention assessments as the experimental group, including tactile sensitivity testing with von Frey monofilaments, the Fugl-Meyer Assessment, the Action Research Arm Test (ARAT), and the Nine-Hole Peg Test (9HPT). This arm serves as a control condition to evaluate the specific effects of the active touch-based sensory intervention on sensory and motor recovery in stroke survivors.

INTERVENTIONS:
Device: Active Touch-Based Sensory Training — This intervention combines functional electrical stimulation with active tactile exploration of virtual textures. Using a touch-sensitive screen and a programmable functional electrical stimulator (MotionStim 8), participants explore two invisible virtual textures by moving their index finger across the screen. Each time the finger crosses a virtual texture line, an electrical pulse is delivered to the finger, simulating tactile sensation. Participants are asked to compare the density of two virtual textures and select the denser one. The stimulation is synchronized with finger movement to ensure real-time sensory feedback. The training consists of 50 trials divided into 5 blocks, and is designed to enhance tactile discrimination and proprioception through sensorimotor integration. The paradigm is interactive, personalized based on individual sensory thresholds, and aims to promote neural plasticity in stroke survivors.
  Arms: Active Touch Sensory Training Intervention

SUMMARY:
Parallel-group, single-blinded controlled clinical trial. The study includes people aged 18-80 years, more than one month after stroke, with confirmed diagnosis, MoCA ≥ 20, and Barthel Index ≥ 3.

The control group receives standard rehabilitation. The experimental group also receives active sensory training with programmable electrical stimulation to simulate virtual textures.

Sensory function was assessed before and after the training using standard tests, including Fugl-Meyer, ARAT, 9HPT, and monofilament testing.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of long-term disability worldwide. In many cases, it results in persistent sensorimotor deficits in the upper limbs, including reduced tactile sensitivity, poor proprioception, and impaired fine motor skills. These deficits limit independence in daily activities such as grasping, dressing, or using utensils, and reduce the quality of life for stroke survivors.

Sensory rehabilitation is a critical but often under-addressed aspect of post-stroke recovery. Traditional approaches frequently focus on motor function alone, overlooking the importance of sensory input in guiding and refining movement. While methods such as sensory stimulation and retraining have shown some promise, their long-term effectiveness remains inconsistent, and they often lack patient engagement.

The present study investigates the efficacy of a novel method of active sensory rehabilitation based on simulated texture exploration using programmable transcutaneous electrical stimulation. This method is designed to combine active tactile exploration with real-time sensory feedback. Participants use their index finger to explore virtual textures on a tablet screen. Each time the finger crosses a virtual texture line, an electrical pulse is delivered to the finger via surface electrodes. This setup creates the sensation of moving across textures of different densities, which the participant must compare and identify.

The goal is to determine whether this approach improves tactile discrimination and supports motor recovery in the upper limb. The trial is conducted as a parallel-group, single-blinded controlled clinical study. Participants are adults aged 18 to 80 years, at least one month post-stroke, with sufficient cognitive and functional status (MoCA ≥ 20, Barthel Index ≥ 3). Participants are randomly assigned to either a control group or an experimental group.

The control group receives conventional rehabilitation prescribed by their physician.

The experimental group receives the same conventional therapy, plus 10 sessions of active sensory training using the programmable stimulation system.

Each session includes 5 blocks of 10 trials, during which the participant explores and compares pairs of virtual textures. Performance data, such as accuracy and response time, are recorded.

Before and after the intervention period, participants are assessed using standard clinical scales: Fugl-Meyer Assessment (FMA) for motor function, Action Research Arm Test (ARAT), Nine-Hole Peg Test (9HPT) for fine motor skills, Touch-Test monofilaments for tactile sensitivity

Results are expected to provide insight into the role of active sensory engagement in neurorehabilitation and help develop more effective strategies for upper limb recovery after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Episode of stroke confirmed by neuroimaging
* More than one month post-stroke
* Montreal Cognitive Assessment (MoCA) score ≥ 20
* Barthel Index score ≥ 3
* Ability to understand and follow instructions
* Informed consent for participation and data collection
* Age 18-80 years

Exclusion Criteria:

* Presence of depressive symptoms (HADS-Depression > 11)
* Upper limb paresis score below 35 on the Fugl-Meyer scale
* Sensory impairment score below 3 or above 10 on the Fugl-Meyer scale

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in Tactile Sensitivity of the Affected Index Finger | From enrollment to the end of treatment at 2 weeks
  Tactile sensitivity is assessed using von Frey monofilaments applied to the index finger of the hand contralateral to the stroke lesion. The outcome is defined as the change in sensory threshold (in grams) from baseline to post-intervention. A decrease in threshold indicates improved tactile sensitivity. This measure evaluates the primary therapeutic effect of the active touch-based sensory training.

SECONDARY OUTCOMES:
Change in Fugl-Meyer Assessment (FMA) Score | From enrollment to the end of treatment at 2 weeks
  To evaluate potential improvements in upper limb motor function following the Active Touch-based sensory training, participants completed the Fugl-Meyer Assessment (FMA) of Sensorimotor Function before and after the intervention. The FMA is a comprehensive scale that measures motor function, sensory function, balance, and joint range of motion in individuals with neurological conditions. The scale's scores range from a minimum of 0 to a maximum of 226, with higher scores indicating a better outcome, reflecting improved motor and sensory function. Scores were compared between the experimental and control groups to assess the effect of the training on motor recovery.
Change in Action Research Arm Test (ARAT) Score | From enrollment to the end of treatment at 2 weeks
  The Action Research Arm Test (ARAT) was used to assess fine and gross motor function of the upper limb. The ARAT is a scale specifically designed to evaluate the ability to perform a range of tasks, including grasp, grip, pinch, and gross movement. The ARAT score ranges from a minimum of 0 to a maximum of 57, with higher scores indicating a better outcome, reflecting improved motor function. Changes in ARAT scores before and after the intervention were analyzed to determine whether sensory training contributed to motor recovery in the experimental group.
Change in Nine-Hole Peg Test (9HPT) Performance | From enrollment to the end of treatment at 2 weeks
  To evaluate changes in manual dexterity, participants performed the Nine-Hole Peg Test at baseline and post-intervention. Task completion time was compared pre- and post-treatment to identify improvements in fine motor skills potentially attributable to the active touch training.

CONTACTS AND LOCATIONS:
Overall Officials: Galina Ivanova, Professor, Study Chair — Federal Center of Cerebrovascular Pathology and Stroke, Russian Federation Ministry of Health
Locations (1):
- Federal Center of Cerebrovascular Pathology and Stroke, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made publicly available, including:
  * Demographic data (age, sex)
  * Clinical characteristics (stroke diagnosis, time since onset)
  * Baseline and post-intervention scores (MoCA, Barthel Index, FMA, ARAT, 9HPT, monofilament testing)
  * Training performance metrics (accuracy, response times). Data will be deposited on the Open Science Framework (OSF) repository to ensure transparency and facilitate secondary analyses.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Beginning immediately after publication with no end date
Access Criteria: Data will be accessible immediately after publication via OSF under a CC-BY 4.0 license, without restrictions. No approval process is required.

REFERENCES:
- [Background] Kapadia N, Moineau B, Popovic MR. Functional Electrical Stimulation Therapy for Retraining Reaching and Grasping After Spinal Cord Injury and Stroke. Front Neurosci. 2020 Jul 9;14:718. doi: 10.3389/fnins.2020.00718. eCollection 2020. PMID 32742254
- [Background] Oh ZH, Liu CH, Hsu CW, Liou TH, Escorpizo R, Chen HC. Mirror therapy combined with neuromuscular electrical stimulation for poststroke lower extremity motor function recovery: a systematic review and meta-analysis. Sci Rep. 2023 Nov 16;13(1):20018. doi: 10.1038/s41598-023-47272-9. PMID 37973838
- [Background] Elbalawy, Y. M., Fahmy, E. M., Taha, S. I., El Sherbini, A. E. H. I., Abdelghany, A. I., & El-Serougy, H. R. (2020). Effect of Sensory Relearning on Sensory and Motor Functions of the Hand in Patients with Carpal Tunnel Syndrome: A Randomized Controlled Clinical Trial. International Journal of Psychosocial Rehabilitation, 24(05).
- [Background] Jerosch-Herold C. Sensory relearning in peripheral nerve disorders of the hand: a web-based survey and delphi consensus method. J Hand Ther. 2011 Oct-Dec;24(4):292-8; quiz 299. doi: 10.1016/j.jht.2011.05.002. Epub 2011 Jul 28. PMID 21798714
- [Background] Sullivan JE, Hurley D, Hedman LD. Afferent stimulation provided by glove electrode during task-specific arm exercise following stroke. Clin Rehabil. 2012 Nov;26(11):1010-20. doi: 10.1177/0269215512442915. Epub 2012 May 4. PMID 22561099
- [Background] Stein J, Hughes R, D'Andrea S, Therrien B, Niemi J, Krebs K, Langone L, Harry J. Stochastic resonance stimulation for upper limb rehabilitation poststroke. Am J Phys Med Rehabil. 2010 Sep;89(9):697-705. doi: 10.1097/PHM.0b013e3181ec9aa8. PMID 20729650
- [Background] Carlsson H, Lindgren I, Rosen B, Bjorkman A, Pessah-Rasmussen H, Brogardh C. Experiences of SENSory Relearning of the UPPer Limb (SENSUPP) after Stroke and Perceived Effects: A Qualitative Study. Int J Environ Res Public Health. 2022 Mar 18;19(6):3636. doi: 10.3390/ijerph19063636. PMID 35329318
- [Background] Carlsson H, Rosen B, Bjorkman A, Pessah-Rasmussen H, Brogardh C. SENSory re-learning of the UPPer limb (SENSUPP) after stroke: development and description of a novel intervention using the TIDieR checklist. Trials. 2021 Jul 5;22(1):430. doi: 10.1186/s13063-021-05375-6. PMID 34225764
- [Background] Carlsson H, Rosen B, Pessah-Rasmussen H, Bjorkman A, Brogardh C. SENSory re-learning of the UPPer limb after stroke (SENSUPP): study protocol for a pilot randomized controlled trial. Trials. 2018 Apr 17;19(1):229. doi: 10.1186/s13063-018-2628-1. PMID 29665842
- [Background] Turville ML, Walker J, Blennerhassett JM, Carey LM. Experiences of Upper Limb Somatosensory Retraining in Persons With Stroke: An Interpretative Phenomenological Analysis. Front Neurosci. 2019 Jul 24;13:756. doi: 10.3389/fnins.2019.00756. eCollection 2019. PMID 31396040
- [Background] Carey L, Macdonell R, Matyas TA. SENSe: Study of the Effectiveness of Neurorehabilitation on Sensation: a randomized controlled trial. Neurorehabil Neural Repair. 2011 May;25(4):304-13. doi: 10.1177/1545968310397705. Epub 2011 Feb 24. PMID 21350049
- [Background] Carlsson H, Gard G, Brogardh C. Upper-limb sensory impairments after stroke: Self-reported experiences of daily life and rehabilitation. J Rehabil Med. 2018 Jan 10;50(1):45-51. doi: 10.2340/16501977-2282. PMID 29068038
- [Background] Carey LM, Matyas TA, Baum C. Effects of Somatosensory Impairment on Participation After Stroke. Am J Occup Ther. 2018 May/Jun;72(3):7203205100p1-7203205100p10. doi: 10.5014/ajot.2018.025114. PMID 29689179
- [Background] Sullivan JE, Hedman LD. Sensory dysfunction following stroke: incidence, significance, examination, and intervention. Top Stroke Rehabil. 2008 May-Jun;15(3):200-17. doi: 10.1310/tsr1503-200. PMID 18647725
- [Background] Kessner SS, Schlemm E, Cheng B, Bingel U, Fiehler J, Gerloff C, Thomalla G. Somatosensory Deficits After Ischemic Stroke. Stroke. 2019 May;50(5):1116-1123. doi: 10.1161/STROKEAHA.118.023750. PMID 30943883
- [Background] Nowak DA, Hermsdorfer J, Topka H. Deficits of predictive grip force control during object manipulation in acute stroke. J Neurol. 2003 Jul;250(7):850-60. doi: 10.1007/s00415-003-1095-z. PMID 12883929